CLINICAL TRIAL: NCT02895204
Title: The Immune-enhancing Effect of Supplementation With Fermented Maillard Reacted Whey Protein in Nondiabetic and Nonobese Subjects
Brief Title: Effect of Fermented Maillard Reacted Whey Protein on Immune Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SU_immune
Record Dates: First submitted 2016-08-30; First posted 2016-09-09 (Estimated); Last update posted 2017-02-13 (Actual); Status verified 2016-09

CONDITIONS: Immune Deficiency
Keywords: Fermented Maillard reacted whey protein; Natural killer cell activity; Immune function; Pre-albumin; Interleukin-12
MeSH Terms: conditions — Immunologic Deficiency Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Test group (F-MRP) (Experimental): Fermented Maillard reacted whey protein (F-MRP) supplementation
  Interventions: Dietary Supplement: Fermented Maillard reacted whey protein (F-MRP)
- Placebo group (Placebo Comparator): Placebo supplementation
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Fermented Maillard reacted whey protein (F-MRP) — 6g of powder containing 4.2g fermented maillard reacted whey protein
  Arms: Test group (F-MRP)
Dietary Supplement: Placebo — 6g of maltodextrin
  Arms: Placebo group

SUMMARY:
To investigate the impact of supplementing fermented Maillard reacted whey protein (F-MRP) on natural killer (NK) cell activity, circulating cytokines and serum protein levels.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled study was conducted on 80 participant without diabetes and obesity. Over a 8-week testing period, the F-MRP group consumed 6 g of powder containing 4.2 g F-MRP each day, whereas the placebo group consumed the same amount with dextrin. NK cell activity (%) was measured based on the ratios of effector cells (E; peripheral blood mononuclear cells, PBMCs) from each participant to target cells (T; K562 cells) at E:T= 10:1, 5:1, 2.5:1, or 1.25:1.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent
* The levels of white blood cells within range 3x10^3/μL~8x10^3/μL
* Males and females
* 20-70 years old
* Without no severe complications

Exclusion Criteria:

* Diabetes
* White blood cell under 3x10^3/μL or over 8x10^3/μL
* Pregnancy or breast-feeding
* Hypersensitivity or disease history for milk protein
* Liver disease, inflammation disease, or severe kidney failure disease
* Cancer, lung disease, leukemia, or autoimmune disease
* Psychological or neurological disease
* Myocardiac infarction or cerebrovascular diseases within 6 months before screening
* Consumption of other test products or drugs within 1 month before screening
* Inflammation related disease within 1 month before screening

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Natural killer cell activity | At baseline
Natural killer cell activity | At 8-week follow-up
Change from baseline natural killer cell activity at 8-week | At baseline and 8-week follow-up

SECONDARY OUTCOMES:
White blood cell | At baseline
White blood cell | At 8-week follow-up
Change from baseline white blood cell at 8-week | At baseline and 8-week follow-up
Interleukin-12 | At baseline
Interleukin-12 | At 8-week follow-up
Change from baseline Interleukin-12 at 8-week | At baseline and 8-week follow-up
Interferon-gamma | At baseline
Interferon-gamma | At 8-week follow-up
Change from baseline Interferon-gamma at 8-week | At baseline and 8-week follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Jong Ho Lee, PhD, Principal Investigator — Yonsei University
Locations (1):
- Yonsei University, Seoul, South Korea